CLINICAL TRIAL: NCT03719456
Title: Prospective Assessment of Procedure-Related and Patient-Reported Outcomes After Retrograde Intrarenal Surgery (RIRS) for Renal Calculi Less Than 20 mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AE 2394
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Renal Stone
Keywords: Renal stone; Calculi; Retrograde Intrarenal Surgery; Flexible ureteroscope
MeSH Terms: conditions — Nephrolithiasis; Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flexible ureteroscope (Experimental)
  Interventions: Procedure: Retrograde Intrarenal Surgery

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery
  Other Names: Flexible ureteroscope

SUMMARY:
The investigators aim at this study to prospectively assess procedure-related outcomes after RIRS for renal calculi less than 20 mm, including stone free rate (SFR), predictors of successful outcome, complications types/rate, readmission rate and the need of auxiliary procedures. In addition, patient-reported outcomes after this modality of intervention are going to be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent.
2. Stone criteria:

   * Less than 20 mm.
   * Infectious stone.
   * Growing stone on follow-up.
3. Kidney criteria:

   * Obstructing stone causing hydronephrosis.
   * Solitary kidney or bilateral renal stones.
4. Patients criteria:

   * Age ≥18 years.
   * Symptomatic stone causing pain or hematuria.
   * Patient comorbidity omitting other modalities as bleeding diathesis or skeletal deformities.
   * Patient preference or patients' social situation concerning profession or amount of travel

Exclusion Criteria:

1. Inability to give informed consent.
2. Stone criteria:

   * More than 20 mm.
   * Peripheral calyceal asymptomatic stone static in size on follow-up.
   * Unsuitable/failure of initial treatment modalities (oral dissolution therapy-SWL) for stones less than 20 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
stone free rate (SFR) | It will be assessed by non contrast computed tomography for the participants one month after the procedure
  stone free rate after the procedure

SECONDARY OUTCOMES:
Predictors of operative time of the procedure | Immediately after the procedure
  Predictors of operative time of the procedure
- Post-operative complications using modified Dindo-Clavian grading system | within 30 days after the procedure
  - Post-operative complications (Type/rate/predictors) using modified Dindo-Clavian grading system
Intra-operative clinical judgment of the surgeon on stone free status using flouroscopy and visual scanning of pelvicalyceal system and its relation to post-operative NCCT. | Post operative day 1 after the procedure
  - Intra-operative surgeon perspective about procedure outcome and its relation to post-operative NCCT.
- Patient -reported outcomes about post operative pain using visual analogue scale | within 3 months after the procedure
  • Post-operative pain: Postoperative pain will be evaluated in all patients by using visual analogue scale (VAS). The impact of patient-related, stone-related and procedure-related factors.
Patient -reported outcomes about General impression on the procedure using Freiburg Index of patient Satisfaction (FIPS). | within 3 months after the procedure
  Patient -reported outcomes about General impression on the procedure using Freiburg Index of patient Satisfaction (FIPS).
Assessment of patient-reported outcomes using patient-reported outcomes measurements information system (PROMIS) | within 3 months after the procedure
  Procedure impact on improvement in patient-reported outcomes measurements information system (PROMIS): PROMIS is a National Institute of Health (NIH) validated system to assess patient quality of life. The PROMIS survey consists of 43 questions assessing the following categories: anxiety/fear, depression/ sadness, fatigue, pain interference, physical function, and sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, MD, Principal Investigator — Urology and Nephrology Center
Locations (2):
- Egypt (2):
  - Urology and Nephrology Center, Al Mansurah, DK
  - Amr A Elsawy, Al Manşūrah

IPD SHARING:
Plan to Share IPD: Undecided